CLINICAL TRIAL: NCT06973304
Title: An Open-label, Phase 3 Study to Evaluate the Efficacy, Safety and Pharmacokinetics of 0.05 mg/kg/Day Subcutaneous Teduglutide Following Treatment of Short Bowel Syndrome for 24 Weeks in Chinese Adults Who Are Dependent on Parenteral Support
Brief Title: A Study of Teduglutide in Chinese Adults With Short Bowel Syndrome
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TAK-633-3009
Record Dates: First submitted 2025-05-08; First posted 2025-05-15 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: Short Bowel Syndrome
Keywords: Drug Therapy
MeSH Terms: conditions — Short Bowel Syndrome | interventions — teduglutide; ALX-0600

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Teduglutide 0.05 milligram per kilogram (mg/kg) (Experimental): Participants will receive teduglutide 0.05 mg/kg subcutaneous (SC) injection, once daily into 1 of the 4 quadrants of the abdomen or either thigh or arm for 24 weeks.
  Interventions: Drug: Teduglutide

INTERVENTIONS:
Drug: Teduglutide — Teduglutide 0.05 mg/kg SC injection.
  Other Names: TAK-633; A16AX08; Revestive; Gattex

SUMMARY:
The main aim of the study is to assess how well teduglutide works over 24 weeks in Chinese adult participants with short bowel syndrome (SBS) who need parenteral support and to see how much it can reduce the amount of parenteral support and understand how the body absorbs, processes, and gets rid of teduglutide.

Participants will receive a daily injection of teduglutide under the skin for 24 weeks. Safety of teduglutide will be checked for 24 weeks after treatment.

Participants will be in the study for about 65 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females 18 years of age or older at the time of signing the informed consent.
2. Intestinal failure due to SBS as a consequence of major intestinal resection (example, due to injury, volvulus, vascular disease, cancer, Crohn's disease).
3. Has undergone intestinal resection resulting in at least 12 continuous months of PS dependency prior to signing the informed consent.
4. Requires PS at least 3 times per week or at least 4 liters per week during the 2 weeks prior to baseline to meet caloric, fluid, or electrolyte needs due to ongoing malabsorption.
5. Has a stable PS requirement for at least 4 consecutive weeks immediately prior to the start of teduglutide treatment. Stability is defined as follows:

   1. Actual PS usage is similar to prescribed PS.
   2. Baseline (Visit 2) 48-hour intake (I)/output (O) volumes should fall within +-25% of the respective 48-hour I/O volumes at the last optimization visit.
   3. The 48-hour urine output volume must not be less than 2 liters and should not exceed 4 liters at the last optimization visit, the stabilization visit, and the baseline visit.
6. Participants with a history of Crohn's disease must be in endoscopic remission for at least 12 weeks prior to the baseline visit.

Exclusion Criteria:

1. Pregnant or lactating female.
2. Participation in a clinical study using an experimental drug within 30 days or 5 half-lives, whichever is longer, prior to screening, or concurrent participation in any other clinical study.
3. Use of glucagon-like peptide (GLP)-2 or human growth hormone or analogs of these hormones within the past 6 months prior to the baseline visit.
4. Use of octreotide, GLP-1 analogs, or dipeptidyl peptidase-4 inhibitors within 30 days prior to the baseline visit.
5. Previous use of teduglutide.
6. Active inflammatory bowel disease (IBD) or any participant with IBD requiring immunosuppressant therapy (example, azathioprine,anti-tumor necrosis factor [anti-TNF]) drugs) that had been introduced or changed within the past 6 months prior to the baseline visit.
7. Intestinal malabsorption due to a genetic condition, such as cystic fibrosis, microvillus inclusion disease, familial adenomatous polyposis.
8. Chronic intestinal pseudo-obstruction or severe dysmotility.
9. Clinically significant intestinal stenosis or obstruction, or evidence of such on upper gastrointestinal (UGI)/small bowel follow-through (SBFT), within the past 6 months prior to the baseline visit.
10. Major gastrointestinal (GI) surgical intervention, including significant intestinal resection, within the past 3 months (insertion of feeding tube, anastomotic ulcer repair, minor intestinal resections less than or equal to [<=] 10 centimeter [cm], or endoscopic procedure is allowed) prior to the baseline visit.
11. Unstable cardiac disease, (example, congestive heart failure, cyanotic disease, or congenital heart disease).
12. Moderate or severe renal impairment, defined as creatinine clearance less than 50 milliliters per minute (mL/min).
13. Currently diagnosed with cancer or a history of any cancer except surgically cured skin cancer within the past 5 years.
14. Severe hepatobiliary disease including any of the following:

    1. Total bilirubin level at least 2 times the upper limit of normal (ULN), except for increased indirect (unconjugated) bilirubin in a patient with Gilbert's syndrome.
    2. AST at least 5*ULN.
    3. ALT at least 5*ULN
15. Active clinically significant pancreatic disease, including clinical signs of pancreatitis associated with elevations in serum amylase or lipase at least 2*ULN.
16. More than 4 SBS-related or PS-related hospital admissions (example, central line-associated bloodstream infection, bowel obstruction, severe fluid/electrolyte disturbances) within the past 12 months prior to the baseline visit.
17. Unscheduled hospitalization within 30 days prior to screening.
18. Non-herpetic viral diseases:

    1. Presence of hepatitis C virus (HCV) antibody and a positive confirmatory test result for HCV RNA (ribonucleic acid) (nucleic acid test or polymerase chain reaction).
    2. Presence of (Hepatitis B Surface Antigen Positive [HBsAg+]). For participants who are negative for HBsAg but are positive for either surface antibodies and/or core antibodies, hepatitis B virus (HBV) deoxyribonucleic acid (DNA) polymerase chain reaction will be performed; if any test result meets or exceeds detection sensitivity, the subject will be excluded.
    3. Positive results for human immunodeficiency virus (HIV) by serology, regardless of viral load.
19. Any condition, disease, illness, or circumstance that in the investigator's opinion puts the participant at any undue risk, prevents completion of the study, or interferes with analysis of the study results. Example of potential disease state/illnesses that may be excluded are listed in the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Estimated)
Dates: Start 2025-06-26 (Actual); Primary Completion 2027-02-10 (Estimated); Study Completion 2027-07-28 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants Who Achieved At Least 20 Percent (%) Reduction From Baseline in Weekly Parenteral Support (PS) Volume at Week 20 and Maintained Through Week 24 | Up to Week 24

SECONDARY OUTCOMES:
Absolute Change From Baseline in Weekly PS Volume up to Week 24 | Baseline up to Week 24
Percent Change From Baseline in Weekly PS Volume up to Week 24 | Baseline up to Week 24
Absolute Change From Baseline in Days Per Week of PS up to Week 24 | Baseline up to Week 24
Percent Change From Baseline in Days Per Week of PS up to Week 24 | Baseline up to Week 24
Number of Participants Who Achieved At Least 20% Reduction From Baseline in Weekly PS Volume at each visit | Up to Week 24
Number of Participants With At Least a 20% Reduction From Baseline in Weekly PS at Week 20 and Maintained Through Week 24 | Baseline, Week 20 and Week 24
Number of Participants With At Least a 2-liter Reduction From Baseline in Weekly PS at Week 20 and Maintained Through Week 24 | Baseline, Week 20 and Week 24
Number of Participants who are able to Completely Wean off of PS support at Week 24 | At Week 24
Time From First Dose to Time of Completely Weaning off of PS Support | Up to Week 24
AUC0-inf: Area Under the Plasma Concentration-time Curve From Time 0 to Time of Infinity for Teduglutide | Predose, 1, 2, 4, 6, 8, and 10 hours post-dose
AUC0-last: Area Under the Plasma Concentration-time Curve From Time 0 to Time of the Last Quantifiable Concentration for Teduglutide | Predose, 1, 2, 4, 6, 8, and 10 hours post-dose
Cmax: Maximum Observed Plasma Concentration for Teduglutide | Predose, 1, 2, 4, 6, 8, and 10 hours post-dose
Tmax: Time to Reach the Cmax for Teduglutide | Predose, 1, 2, 4, 6, 8, and 10 hours post-dose
T1/2: Terminal Phase Half-life for Teduglutide | Predose, 1, 2, 4, 6, 8, and 10 hours post-dose
CL/F: Apparent Clearance for Teduglutide | Predose, 1, 2, 4, 6, 8, and 10 hours post-dose
V/F: Apparent Volume of Distribution During the Terminal Elimination Phase for Teduglutide | Predose, 1, 2, 4, 6, 8, and 10 hours post-dose
Plasma Concentrations of Teduglutide | At Week 4 and Week 24
Number of Participants With Positive Antidrug Antibodies (Neutralizing and Non-neutralizing) | Baseline, Week 4, and Week 24
Number of Participants Who Experienced At Least One Treatment-emergent Adverse Event (TEAE), Serious Adverse Event (SAE), and Adverse Event of Special Interest (AESI) | From first dose of study drug up to follow-up (Week 48)
Change From Baseline in 48-hour Urine Output | Baseline up to 48 hours
Change From Baseline in Body Weight | Baseline up to Week 48
Change From Baseline in Body Mass Index | Baseline up to Week 48

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (4):
- China (4):
  - Beijing Tsinghua Changgung Hospital, Changping, Beijing Municipality
  - Peking Union Medical College Hospital, Dongcheng, Beijing Municipality
  - Affiliated Jinling Hospital, Medical School of Nanjing University, Nanjing, Jiangsu
  - Zhongshan Hospital, Xiamen University, Siming, Xiamen

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: Click here for more information about this trial in easy-to-understand language, including a Plain Language Summary of the results if the trial has been completed. — https://clinicaltrials.takeda.com/study-detail/579550b2ccf649ac??page=1&idFilter=TAK-633-3009